CLINICAL TRIAL: NCT07020390
Title: The Effect of Anesthesia Techniques on Quality of Recovery (QoR-40) Scores in Benign Prostatic Hyperplasia (Holmium Laser Enucleation of the Prostate - HoLEP) Surgery: A Cross-Sectional, Observational, Prospective Study
Brief Title: Effect of Anesthesia Techniques on Quality of Recovery Scores in HOLEP Surgery
Status: Recruiting | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gamze Talih, Principal Investigator, TC Erciyes University
Other Study IDs: 2025/195
Record Dates: First submitted 2025-06-03; First posted 2025-06-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-06

CONDITIONS: HoLEP; QoR-40; Anesthesia, General; Anesthesia,Spinal; Anesthesia; Combine Spinal and Epidural
Keywords: HoLEP; Quality of recovery (QoR-40); Patient satisfaction; Spinal anesthesia; General anesthesia; Benign prostatic hyperplasia; spinal-epidural anesthesia
MeSH Terms: conditions — Patient Satisfaction; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who undergoing HOLEP under different anesthesia methods
  Interventions: Procedure: Anesthesia method

INTERVENTIONS:
Procedure: Anesthesia method — Patients will be divided into subgroups according to different anesthesia methods (general, spinal, and combined spinal-epidural anesthesia) and compared in terms of recovery quality (QoR-40) and other parameters.

SUMMARY:
The aim of this observational study is to evaluate the effects of different anesthesia techniques on the quality of recovery (QoR) and patient satisfaction in male patients, typically older adults with benign prostatic hyperplasia, undergoing Holmium Laser Enucleation of the Prostate (HoLEP).

Participants will undergo HoLEP surgery under one of three anesthesia techniques-general, spinal, or combined spinal-epidural anesthesia-and will complete the QoR-40 questionnaire both before and after the surgery.

DETAILED DESCRIPTION:
These patients will be informed about the preoperative study and the Quality of Recovery 40 (QoR-40) scoring scale will be applied by the responsible researcher preoperatively and within 24 hours postoperatively, and the values will be recorded. The anesthesia method of the patients will be determined as determined routinely according to the patient's age, additional diseases, duration of surgery, and patient preference and will be applied by an experienced anesthesiologist. Routine intraoperative follow-ups of all patients will be performed. Surgeries completed without any complications will be taken to the recovery unit at the end of the procedure, and stable patients will be transferred to the ward. In patients whose ward follow-ups continue routinely, catheter-related bladder discomfort will be evaluated within 24 hours postoperatively, postoperative patient and surgeon satisfaction will be evaluated according to the 5-point Likert scale, and the QoR-40 score will be recorded. Postoperative pain levels and analgesic needs will be recorded. Parameters will be compared by dividing into groups according to the anesthesia method.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for HOLEP surgery due to benign prostatic hyperplasia.
* Patients who consent to participate in the study.

Exclusion Criteria:

* Refusal to participate in the study
* Presence of cognitive impairment
* Use of psychoactive medications
* Failure of the intraoperative anesthesia technique and necessity to change the anesthesia method
* Requirement for reoperation or admission to the intensive care unit
* Voluntary withdrawal from the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals have biologically male anatomy relevant to the procedure are eligible to participate.
Study Population: Patients aged 18 years or older who meet the eligibility criteria and are scheduled to undergo surgery for benign prostatic hyperplasia (BPH).
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
The Quality of Recovery Score (QoR-40) | Baseline (preoperative) and postoperative day 1
  The QoR-40 is a self-rated questionnaire that consists of 40 items to evaluate the pain levels and physical and emotional state of patients, comprising five subscales: emotional state (n = 9), physical comfort (n = 12), patient support (n = 7), physical independence (n = 5), and pain (n = 7). Each item is scored on a five-point Likert scale ranging from 1 to 5. The scores for the subscales are given by the sum of the corresponding items, and the total score is computed by a summation of all items. The total score ranges from 40 to 200. Higher scores indicate higher levels of functioning or well-being.
  Change in QoR-40 score from preoperative to postoperative day 1 to evaluate overall recovery quality.

SECONDARY OUTCOMES:
Patient satisfaction and surgeon satisfaction | Postoperative day 1
  Patient and surgeon satisfaction was rated using a 5-option Likert scale at postoperative day 1: 1 = very bad, 2 = bad, 3 = moderate, 4 = good and 5 = excellent.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Melikgazi, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No